CLINICAL TRIAL: NCT02932241
Title: Computerized DBT Skills Training for Suicidal and Heavy Episodic Drinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Chelsey Wilks, Graduate Student, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002445; F31AA024658-01 (NIH)
Record Dates: First submitted 2016-10-10; First posted 2016-10-13 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Suicidal Ideation; Alcohol Drinking
MeSH Terms: conditions — Suicidal Ideation; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computerized DBT skills training (Experimental): The Computerized Dialectical Behavior Therapy Skills Training (cDBT) intervention includes 4 mindfulness, 6 emotion regulations, 2 distress tolerance, and 4 addiction skills. cDBT will retain the essence of DBT skills by being didactically focused, having a predetermined agenda driven by skills to be taught, emphasizing modeling through video vignettes, incorporating in session practice of skills whenever feasible, reviewing homework at beginning of sessions before teaching new skills, and assigning practice between sessions.
  Interventions: Behavioral: Computerized Dialectical Behavior Therapy Skills Training
- Waitlist (No Intervention): A waitlist (WL) control condition was chosen considering the pilot nature of the study, feasibility, and the overall goal of assessing treatment's promise. Participants will be assessed for drinking and suicidal urges in the same manner as in the cDBT condition. After 8 weeks, subjects will be able to enroll in the intervention.

INTERVENTIONS:
Behavioral: Computerized Dialectical Behavior Therapy Skills Training — 8, 50 minute skill training sessions made available to participants each week
  Arms: Computerized DBT skills training

SUMMARY:
Alcohol use is considered to be a significant risk factor among those who die by suicide, especially among those who drink to regulate their emotions. Unfortunately, there is a dearth of treatment outcome research for suicidal heavy drinkers. Further, treatments that target this population must be maximally effective, with promise for wide dissemination. The application of technology has been increasingly utilized as an efficacious and acceptable way to rapidly disseminate evidence-base treatment. However, these methods are used infrequently for individuals deemed too high risk for computerized treatment. Along these lines, the goal of this project is to begin a line of research focused on developing interventions to reduce heavy drinking and risk for suicide through the use of technology. Dialectical Behavior Therapy (DBT) skills training is an effective intervention for behaviors associated with emotion dysregulation including addictive and suicidal behaviors. Further, DBT skills use has been identified as the active ingredient for treatment effectiveness; thus, a skills training intervention delivered via the Internet has the capacity to be a potent and efficient method of treatment delivery. The goal of this research is to establish a proof of concept for developing and evaluating a potentially efficacious and acceptable intervention for heavy episodic drinkers who are suicidal. Specifically, this project proposes to conduct a randomized controlled pilot trial of a computerized DBT skills training intervention for suicidal individuals who engage in heavy episodic drinking (HED) to regulate emotions. The project's aims are to conduct a randomized controlled pilot trial of cDBT vs. a Wait-list control (WL). This pilot trial is not intended to demonstrate that cDBT works better than other interventions in improving clinical indices, but rather to determine whether further revisions of the cDBT intervention are needed and will inform the design of a subsequent full-scale randomized controlled trial.

DETAILED DESCRIPTION:
It is well established that clinical research should focus on streamlining treatments in ways that maximizes their potency and ease of implementation. The application of technology has been increasingly utilized as an effective and acceptable way to rapidly disseminate evidence-base treatment. However, these methods are used infrequently for individuals deemed too high risk for computerized psychotherapy. This atheoretical approach to participant exclusion broadens the treatment gap among those in dire need of treatment. Along these lines, the primary goal of this project is to establish a proof of concept for developing and evaluating an efficacious and acceptable intervention for heavy episodic drinkers who are suicidal.

This scope has been selected to increase feasibility for this pilot trial and to allow comparison with a wait-list control condition, providing important groundwork for a subsequent randomized control trial. The proposed research will take place in one phase and will fall within Stage 1a and 1b of the updated Stage Model for Behavioral Therapy Research. This project will consist of a randomized controlled pilot trial, an initial "strong test" of efficacy of cDBT for the treatment of HED and suicidal behaviors, using a between groups design. This method of intervention delivery (e.g. computerization) will allow for ease of transition to subsequent stages that fit the updated scope of Behavioral Therapy Research which highlight the need for dissemination and implementation. The overall aim of this project is not to demonstrate that cDBT works better than other interventions in improving outcomes, but rather to provide preliminary evidence that the intervention is feasible and efficacious in producing change when delivered through an easily disseminated and acceptable method.

The primary goal of computerized DBT Skills Training will be to eliminate HED and suicidal behavior that function to regulate emotions while simultaneously increasing behavioral control through the use of functional, skillful behavior. cDBT-ER is an existing 8-week computerized skills intervention that targets difficulties in emotion regulation and includes numerous skills that explicitly target modifying emotional states. DBT skills translate well into computerized interventions, as they are based on learning models in which patients are taught reproducible skills to be used in their environment. The proposed intervention will require adding the DBT addiction skills to target heavy drinking as well as including a computerized version of a risk assessment protocol to assess suicidal urges electronically. The DBT addiction skills draw largely from relapse prevention and include DBT adaptations of Harm Reduction (via "Dialectical Abstinence") and Urge Surfing (via "Burning Bridges). The addiction skills have been implemented in numerous DBT studies that explicitly target addictive behavior with positive outcomes in reducing substance and alcohol use. Thus, cDBT would teach clients ways to reduce and eliminate alcohol consumption, along with skillful behaviors to effectively manage negative emotions.

ELIGIBILITY:
Inclusion Criteria:

1. Current suicidal ideation in last 4 weeks
2. Heavy episodic drinkers (reporting consumption of 4 drinks for women and 5 drinks for men over a 2 hour period at least twice in the past month)
3. High emotion dysregulation defined as being one standard deviation above the mean on the DERS
4. Age >=18 years old
5. English speaking
6. Medication usage stabilized
7. Consents to study
8. Has Internet & phone access

Exclusion Criteria:

1. Bipolar I, Schizophrenia, Schizophreniform, Schizoaffective Disorders, Psychosis,
2. Lives outside of referral network (U.S).
3. Court ordered for treatment
4. Unable to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Alcohol Use | 16 weeks
  Time line follow back to assess quantity and frequency

SECONDARY OUTCOMES:
Acceptability, as measured by the Client Satisfaction Inventory (CSI). | 8 weeks
  The degree to which this population experiences satisfaction with the intervention.
Suicidal ideation, as measured by the Beck's Scale for Suicidal Ideation (BSSI). | 16 weeks
  Severity of suicidal ideation.

CONTACTS AND LOCATIONS:
Overall Officials: Chelsey R Wilks, M.S., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have yet to determine whether or not to share data; if so, all data would be de-identified.

REFERENCES:
- [Derived] Yin Q, Wilks CR. Untangling the temporal association between daily urges to die by suicide and to use substances. Psychiatry Res. 2023 May;323:115178. doi: 10.1016/j.psychres.2023.115178. Epub 2023 Mar 22. PMID 37012190
- [Derived] Wilks C, Yin Q, Ang SY, Matsumiya B, Lungu A, Linehan M. Internet-Delivered Dialectical Behavioral Therapy Skills Training for Suicidal and Heavy Episodic Drinkers: Protocol and Preliminary Results of a Randomized Controlled Trial. JMIR Res Protoc. 2017 Oct 25;6(10):e207. doi: 10.2196/resprot.7767. PMID 29070480